CLINICAL TRIAL: NCT00772837
Title: Effect of Eradication of Helicobacter Pylori on the Dyspeptic Symptoms.
Acronym: EEHPDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: DR.SHAHAB ABID, SECTION OF GASTROENTEROLY,DEPARTMENT OF MEDICINE,AGA KHAN UNIVERSITY
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 602-Med/ERC-06
Record Dates: First submitted 2008-10-14; First posted 2008-10-15 (Estimated); Last update posted 2009-11-10 (Estimated); Status verified 2009-11

CONDITIONS: Functional Dyspepsia; Helicobacter Pylori Infection
Keywords: Functional Dyspepsia; Helicobacter Pylori eradication; Quality of Life; Dyspeptic Symptoms
MeSH Terms: interventions — Omeprazole; Clarithromycin; Amoxicillin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1.H.Pylori Eradication Group (Experimental): The eradication group will receive triple therapy (omeprazole 20mg BID for 1 week along with Clarithromycin 500mg BID and Amoxycillin 1g BID) for 1 week for the eradication of H. pylori
  Interventions: Drug: Omeprazole + Clarithromycin + Amoxycillin
- 2.Control Placebo Group (Placebo Comparator): The control group will receive omeprazole 20 mg BID for 1 week along with placebo antibiotics for 1 week
  Interventions: Drug: Omeprazole + placebo antibiotics

INTERVENTIONS:
Drug: Omeprazole + Clarithromycin + Amoxycillin — Omeprazole 20mg BID for 1 week along with Clarithromycin 500mg BD and Amoxycillin 1g BD for 1 week
  Arms: 1.H.Pylori Eradication Group
Drug: Omeprazole + placebo antibiotics — omeprazole 20 mg bid for 1 week along with placebo antibiotics for 1 week
  Arms: 2.Control Placebo Group

SUMMARY:
Helicobacter pylori eradication and its impact on symptoms in patients with non-ulcer dyspepsia remain controversial . Many studies have examined the effect of H. pylori eradication on dyspeptic symptoms, but the results have been conflicting and inconclusive, with as many studies yielding positive as negative results. Some studies have shown a significant (although weak) symptomatic improvement after H. pylori eradication, and while other yielding negative results. A recent Cochrane review has comprehensively demonstrated that H.pylori eradication therapy has a small but statistically significant effect in H.pylori positive non-ulcer dyspepsia. An economic model suggests this modest benefit may still be cost effective . However it is difficult to reconcile these results in areas with very high prevalence of H. pylori infection such as Pakistan since no such studies have been conducted in developing countries.

The investigators hypothesize that eradication of Helicobacter pylori (H. pylori) leads to a sustained improvement in symptoms of patients diagnosed with H. pylori associated functional (non-ulcer) dyspepsia.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory adult males and non-pregnant females.
* Dyspeptic symptoms for at least 3 months.
* Normal endoscopic findings.
* H. Pylori positive on testing.

Exclusion Criteria:

* Patients with erosive and non erosive esophagitis.
* Barrette's esophagus.
* Duodenal Ulcer, Gastric Ulcer or gastric erosions.
* Patients with known sensitivity to antibiotics.
* Patients with severe concomitant systemic disease.
* Patients with upper GI surgery except cholecystectomy.
* Females with pregnancy or breast-feeding.
* Malignancy
* Alarm symptoms such as bleeding per rectum, hematemesis, and severe weight loss.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Actual)
Dates: Start 2006-08; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Improvement in Dyspeptic Symptoms after eradication of Helicobacter Pylori in Patients with Functional Dyspepsia | 1 year

SECONDARY OUTCOMES:
To determine whether eradication of Helicobacter Pylori improves the quality of life in patients with Functional Dyspepsia i.Quality of life (QoL) assessment on the basis of SF-36. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: DR.SHAHAB ABID, MD, Principal Investigator — Aga Khan University
Locations (1):
- Aga khan University, Karachi, Sindh, Pakistan